CLINICAL TRIAL: NCT04207762
Title: Evaluation of the Safety and Sensitivity of 18F-AmBF3-TATE PET/CT for Imaging NET Patients
Brief Title: 18F-AmBF3-TATE PET/CT for Imaging NET Patients
Status: Completed | Type: Observational
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Other Study IDs: H19-03674
Record Dates: First submitted 2019-12-16; First posted 2019-12-23 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2019-12

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PET/CT Diagnostic Imaging: Each subject will have a PET/CT scan, using 18F-AmBF3-TATE. 18F-AmBF3-TATE radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada.
  Interventions: Diagnostic Test: 18F-AmBF3-TATE PET/CT; Diagnostic Test: Routine blood draw

INTERVENTIONS:
Diagnostic Test: 18F-AmBF3-TATE PET/CT — Blood pressure, heart rate, and oxygen saturation levels and EKG monitoring (vital signs) will be recorded prior to the injection and at three other stages of the scan visit. Each study subject will have an intravenous catheter inserted. Prior to the radiotracer injection an ultra low dose CT will be taken. Subjects are positioned supine, arms down. The subject will receive a bolus intravenous dose of the radiotracer from an approved study supplier site. A Dynamic PET scan will be taken of the heart. Then a serial whole body PET scan will be done. Vital signs will be taken again and the subject will have a bathroom break. The patient will return to the scanner bed for a standard low dose CT and whole body PET scan. Vital signs will be taken again, and subject will be allowed to use the washroom again. The subject will return to the scanner bed for the final time for an ultra low dose CT and whole body PET scan. A final set of vitals will be taken and the subject will be discharged.
Diagnostic Test: Routine blood draw — Complete blood counts and routine clinical chemistry performed before and repeated within 18-72 hours after [18F]AmBF3-TATE administration.

SUMMARY:
Neuroendocrine tumours (NETs) are generally slow growing, but some can be aggressive and resistant to treatment. Compared to healthy cells, the surface of these tumor cells has a greater number of special molecules called somatostatin receptors (SSTR). Somatostatin receptor scintigraphy and conventional imaging are used to detect NETs.

This study proposes 18F-AmBF3-TATE positron emission tomography/computed tomography (PET/CT) is superior to current imaging techniques. The goal is to evaluate the biodistribution and safety of 18F-AmBF3-TATE PET/CT for neuroendocrine tumour imaging.

DETAILED DESCRIPTION:
Each subject will have a PET/CT scan using 18F-AmBF3-TATE. The 18F-AmBF3-TATE radioactive tracer is manufactured for this study under a Clinical Trial Application filed with Health Canada.

After providing informed written consent subjects will complete a medical history questionnaire.

Monitoring of adverse events There will be short-term evaluation of adverse events by comparison of vital signs before and after administration of 18F-AmBF3-TATE . Eighteen to seventy-two hours after 18F-AmBF3-TATE administration the participant will return to the imaging department to perform a follow up safety assessment and routine blood draw. The study coordinator will ask the participant if they have experienced any adverse events during that time period and complete the adverse event questionnaire.

Follow-up Assessments

The following information will be collected up to 12 months following the PET/CT scans:

Initiation of a new treatment, Laboratory results and pathology reports, Results of imaging studies, Final clinical diagnosis by physician and relevant clinical notes. The study is expected to take up to 1 year for accrual.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Participants with newly diagnosed or documented neuroendocrine tumours (NET), with at least one measurable lesion based on CT, MR or at least one visualised lesion on PET/CT imaging (either from an 18F-FDG, 18F-FDOPA or 68Ga-DOTATOC/DOTATATE scan) or scintigraphy (with 111In-pentetreotide imaging).
* ECOG performance status of 2 or less.

Exclusion Criteria:

* Pregnancy
* Medically unstable (eg. acute illness, unstable vital signs)
* Unable to lie supine for the duration of imaging
* Unable to provide written consent
* Exceeds safe weight limit of the PET/CT bed (204.5 kg) or unable to fit through the PET/CT bore (diameter 70 cm)
* Patients with widespread liver metastases occupying more than 50% of the liver volume will not be eligible to participate in this study as this would preclude assessment of normal liver activity for dosimetry purposes.
* Patients with baseline ALT or AST higher than 5× ULN or 250 U/L.
* Patients with elevated baseline levels of total bilirubin (higher than 1.2× ULN, or 1.3 mg/dL, (with exception of Gilbert's syndrome), with INR >1.2, or platelet count below the lower limit of normal (typically <150 000/μL.
* Patients with elevated alkaline phosphatase (ALP), equal to or higher than 2× ULN or 250 U/L, unless the ALP elevation is not from a hepatic origin.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective, open-label trial in patients with proven/documented SSTR positive tumors.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2020-09-21 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Biodistribution of 18F-AmBF3-TATE PET/CT in human subjects | 1 year
  Measurement of radiotracer uptake at multiple time points following radiotracer injection. Calculation of radiation dosimetry using OLINDA 2.0 methodology. Determination of tumour uptake in terms of standardized uptake values and tumour/blood, tumour/liver and tumour/lung ratios (descriptive analysis). For accuracy determination, it is anticipated that only a subset of participants may have a complete gold standard for the determination of accuracy. The sensitivity, specificity and accuracy (along with the confidence interval) of 18F-AMBF3-TATE will be calculated for patients with an available gold standard. The proportion of participants with a complete gold standard is not yet known for this study.

SECONDARY OUTCOMES:
Number of participants with 18F-AmBF3-TATE - related adverse events as assessed by abnormal vital sign measurement. | Before injection, 1 hours post injection, 2 hours post injection and 2.5 hours post injection
  Vital signs (blood pressure, heart rate and pulse oximetry) will be measured at four time points. All values that fall outside of the normal parameters will be assessed by a physician and reported as an adverse event.
Number of participants with self-reported 18F-AmBF3-TATE -related adverse event | 18-72 hours
  Patients will return to the department 18-72 hours after the 18F-AmBF3-TATE PET/CT scan to see if they experienced any adverse events. These are recorded and evaluated for severity and likelihood they are related to the study drug. All adverse events will be recorded and summarized in the final report.
Total number of lesions per anatomic location identified by 18F-AmBF3-TATE PET/CT | 1 year
  All lesions will be tabulated and classified by compartment (pancreas, liver, bowel, lung and mediastinum, abdomen and retroperitoneal lymph nodes, bone, other) for all imaging that has been done for that subject. A total number of lesions will be calculated and a proportion of lesions detected will be reported and will be compared by calculating the median and its confidence interval. This will assess the biodistribution of 18F-AmBF3-TATE PET/CT.

CONTACTS AND LOCATIONS:
Locations (1):
- BC Cancer, Vancouver, British Columbia, Canada